CLINICAL TRIAL: NCT03958175
Title: Screening for Reading Difficulties in Parkinson's Disease: An Evaluation of the Alouette Test
Brief Title: The Alouette Test in Parkinson Disease
Acronym: REPEAT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: REPEAT
Record Dates: First submitted 2019-05-20; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's Disease: Patients with Parkinson's Disease (PD) were evaluated for reading disorders using a screening method validated for dyslexia.
  Interventions: Other: Alouette test (reading test)
- Patients without Parkinson's Disease = control group: Patients without Parkinson's Disease (PD) were evaluated for reading disorders using a screening method validated for dyslexia.
  Interventions: Other: Alouette test (reading test)

INTERVENTIONS:
Other: Alouette test (reading test) — The alouette test was assessed at a fixed distance of 40 centimeters on a fixed surface to avoid errors related to hand tremors.

SUMMARY:
Reading disorders in Parkinson's Disease (PD) are poorly evaluated due to the lack of validated tests to screen for them. They are often attributed to hand tremors associated with the disease. In this study, the investigating team evaluated the "alouette test" validated for dyslexia screening, in PD by comparing the results to healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease
* Montreal Cognitive Assessment (MoCA) test > 20

Exclusion Criteria:

* Patient's with supranuclear Palsy
* Other neurologic disease
* Any ophthalmologic disease
* Presence of a nystagmus
* Visual acuity < 0.6

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Score on the Alouette test | 1 day
  The Alouette test is based on the precision and speed in reading a short text (279 words). The score corresponds to the total number of words correctly read.

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Mathis, Dr, Principal Investigator — Hospices Civils de Lyon